CLINICAL TRIAL: NCT02066662
Title: Influence of Rivaroxaban Compared to Vitamin K Antagonist Treatment Upon Development of Cardiovascular Calcification in Patients With Atrial Fibrillation and/ or Pulmonary Embolism (IRIVASC- Trial)
Brief Title: Rivaroxaban Compared to Vitamin K Antagonist Upon Development of Cardiovascular Calcification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-001
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation or Pulmonary Embolism; Need of Long Term Oral Anticoagulation Therapy (OAT); Existent Coronary or Valvular Calcification, or Both and Agatston Score > 50 in at Least One Location
Keywords: Coronary or Valvular Calcification; Agatston Score; Rivaroxaban; Coumarin; Oral Anticoagulation Therapy (OAT); Atrial Fibrillation; Pulmonary Embolism
MeSH Terms: conditions — Atrial Fibrillation; Pulmonary Embolism | interventions — Rivaroxaban; Phenprocoumon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivaroxaban (Experimental): Arm A: Rivaroxaban (tablet) for patients with atrial fibrillation: with 20 mg once daily for patients with eGFR > 49 ml per minute and 15 mg rivaroxaban once daily for patients with eGFR of 15 to 49 ml. Rivaroxaban (tablet) for patients with pulmonary embolism : 2x a day 15 mg at day 1-21 and 1x 20 mg from day 22 ongoing
  Interventions: Drug: Rivaroxaban or Marcumar
- Marcumar (Active Comparator): Arm B: Adjusted dose coumadin/phenprocoumon (tablet) titrated according to target international normalized ratio (INR) with a target range 2.0 to 3.0.
  Interventions: Drug: Rivaroxaban or Marcumar

INTERVENTIONS:
Drug: Rivaroxaban or Marcumar — Arm A: Rivaroxaban (tablet) for patients with atrial fibrillation: with 20 mg once daily for patients with eGFR > 49 ml per minute and 15 mg rivaroxaban once daily for patients with eGFR of 15 to 49 ml. Rivaroxaban (tablet) for patients with pulmonary embolism : 2x a day 15 mg at day 1-21 and 1x 20 mg from day 22 ongoing;
  Arm B: Adjusted dose coumadin/phenprocoumon (tablet) titrated according to target international normalized ratio (INR) with a target range 2.0 to 3.0.
  Other Names: Xarelto; Marcumar

SUMMARY:
The following trial hypothesis will be proved: In patients with atrial fibrillation and/ or pulmonary embolism standard anticoagulant treatment with coumadin/phenprocoumon is associated with accelerated coronary or valvular calcification as assessed by cardiac computed tomography compared to the new anticoagulant therapy with rivaroxaban.

DETAILED DESCRIPTION:
A multi center, prospective, controlled, open, randomized, interventional clinical trial blinded concerning outcome measurements with a two- arm parallel group design will be performed to investigate the association of rivaroxaban compared to coumadin/phenprocoumon treatment for OAT in patients with atrial fibrillation and / or pulmonary embolism regarding the development and progression of coronary artery calcification (CAC) and aortic valve calcification (AVC) as assessed by multi-slice spiral computed tomography scanning (MSCT) within one year follow-up.

In total 190 patients (95 patients per treatment arm) with atrial fibrillation and/ or pulmonary embolism with the indication for oral anticoagulation therapy will be enrolled.

After screening first cardiac CT scan will be performed in order to validate if calcium score is >50 which is an inclusion criteria. If the patient matches all other inclusion/exclusion criteria the remaining imaging procedures (Echocardiography, Intima Media Thickness of carotid artery (IMT) and Flow Mediated Vasodilatation (FMD), Electrocardiography (ECG) and blood pressure are executed. Pregnancy strip test will be executed and also serum chemistry, hematology, coagulation and batch analysis will be performed.

Patients will then be randomized to one of the two arms (Rivaroxaban or Marcumar) and will undergo the same examinations and measurements as described above at 1 week, 1, 6, 9 and 12 month Follow- Up (FU). In case of a positive result in respect to the primary endpoint a FU after 2 years will be performed.

Primary outcome measures will be assessed after all active patients will have completed 12-months study visit (interim analysis)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged > 18 years
2. Need for long-term OAT according to current international guidelines for the treatment of atrial fibrillation (ACC/(American Heart Association [AHA]/ European Society of Cardiology [ESC]guidelines) and / or pulmonary embolism (ACCP/ESC guidelines).
3. Existent Coronary or Valvular Calcification, or both and an Agatston Score > 50 in at least one location as assessed by MSCT at Screening
4. The anticipated minimum life expectancy is18 months

Exclusion Criteria:

1. Patient has any clinical condition which does not allow initiation of long-term OAT including all contraindications such as hypersensitivity to active ingredient or other excipients, clinically relevant acute bleedings and all other risk circumstances according to Summary of Medicinal Product (SmPC) in which all warnings and preventive measures and precautions are described and have to be kept.
2. Hypersensitivity to active substances investigated or to any of the excipients
3. Patients had a previous coronary stent implantation in a way which makes coronary artery calcification scoring impossible or unreliable and no Valvular Calcification with Agatston Score > 50
4. Chronic kidney disease (CKD) Stage V (GFR <15 mL)
5. Liver disease with coagulopathy or other bleeding disorders including cirrhotic patients with Child Pugh B and C
6. Acute gastrointestinal diseases
7. Clinically significant active bleeding
8. Alcohol, opioids or drug abuse
9. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
10. Patient is unwilling or unable to give informed consent
11. Patient is unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
12. Participation in a parallel interventional clinical trial
13. Patient has been committed to an institution by legal or regulatory order
14. Pregnant or lactating women
15. Female patient capable of bearing children without highly effective methods of birth control
16. Patient receives concomitant treatment with strong concurrent Cytochrome P 450 3A4 (CYP3A4)- and P- glycoprotein (P-gp)- inhibitors, i.e. azole-antimycotics (ketoconazole, itraconazole) or human immunodeficiency virus (HIV) protease inhibitors
17. Neuraxial Anaesthesia or spinal/epidural puncture
18. Known Endocarditis
19. Known Lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-07; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Progression of coronary and aortic valve calcification (Agatston, volume & mass score as assessed by cardiac CT) | Cardiac Computertomography (CT) will be performed at screening, after 12 months and at 24 months
  To investigate the association of rivaroxaban compared to coumadin/phenprocoumon treatment for OAT in patients with atrial fibrillation and / or pulmonary embolism regarding the development and progression of coronary artery calcification (CAC) and aortic valve calcification (AVC) as assessed by multi-slice spiral computed. tomography scanning (MSCT) within one year follow-up

SECONDARY OUTCOMES:
Serum chemistry including Matrix Gla Protein (MPG) level changes and Fetuin-A (baseline/ follow up) | baseline and 12 month Follow Up
Changes in intima-media thickness of carotid artery (IMT) and flow-mediated vasodilation of brachial artery (FMD) | Baseline, 6, 12 and 24 month FU
Progression of aortic calcification (aortic Agatston Score) | screening and 12 month FU
Changes in ventricular diastolic function parameters as determined by echocardiography (strain/strain-rate imaging) | baseline, 6, 9, 12 and 24 month FU

OTHER OUTCOMES:
Occurrence of major cardiovascular complications (MACE) | 1 week, 1, 6, 9, 12 and 24 month FU
Non- major bleedings | 1week, 1, 6, 9, 12 and 24 month FU
Major bleedings | 1 week, 6, 9, 12 and 24 month FU

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Hospital Coburg, Med. Clinic II for Internal Medicine and Cardiology, Coburg, Bavaria
  - University Hospital Aachen, Department of Cardiology, Aachen, North Rhine-Westphalia
  - St.-Antonius-Hospital Eschweiler, Internal Medicine, Eschweiler, North Rhine-Westphalia